CLINICAL TRIAL: NCT05354947
Title: Effects of Multi-Site Abdominal Ultrasound Stimulation on Glycemic Control in T2DM
Brief Title: Ultrasound Effects on Glycemic Control in T2DM
Acronym: U/S_in_T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000032493
Record Dates: First submitted 2022-04-05; First posted 2022-05-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 30 minute, dual site stimulation (Experimental): Ultrasound Deliveryfor 30 minutes total: 15 minutes on the liver target site and 15 minutes on the intestinal target site.
  Interventions: Device: Ultrasound Delivery
- 60 minute, dual site stimulation (Experimental): Ultrasound Delivery for 60 minutes total: 30 minutes on the liver target site and 30 minutes on the intestinal target site.
  Interventions: Device: Ultrasound Delivery

INTERVENTIONS:
Device: Ultrasound Delivery — A General Electric LOGIQ E10 ultrasound machine with a C1-6-XD clear probe, will be used to selectively deliver pulsed ultrasound to both, the portal region of the liver and the superior mesenteric plexus.

SUMMARY:
This is an open label, exploratory pilot study that will assess the effects of dual site focused pulsed ultrasound treatment on glycemic parameters in subjects with T2DM.

DETAILED DESCRIPTION:
This study will test whether multi-site abdominal ultrasound stimulation can have lasting effects on elevated glucose levels in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with a diagnosis of type 2 diabetes ≥ 3 months.
2. Age ≥ 21 and ≤ 75 years.
3. Currently on a stable treatment regimen of oral anti-diabetic drugs and not currently prescribed for medication escalation. Oral anti-diabetic drugs are limited to one or more of the following:

   * Metformin
   * Sulfonylureas
   * Meglitinides
   * Thiazolidinediones
4. HbA1c > 7.0% and < 10% by local laboratory analysis.
5. Body Mass Index (BMI) ≥ 18 to ≤ 40.0 kg/m2.
6. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Principal Investigator.
7. Female subjects must be non-pregnant and non-lactating and have a negative serum pregnancy test at screening and before the ultrasound session.
8. Ability to provide written informed consent.

Exclusion Criteria:

1. History or current diagnosis with T1DM or T2DM subjects on insulin, DPP-4 inhibitors, GLP agonists.
2. A subject who is already indicated for medication escalation of their current diabetic therapy.
3. A subject who has manifestations of advanced complications from poorly controlled or longstanding diabetes such as diabetic retinopathy, diabetic neuropathy and cardiovascular complications including, but not limited to coronary artery disease, peripheral vascular disease, or cerebrovascular disease such as transient ischemic attack [TIA], cerebral infarct, or cerebral hemorrhage.
4. History or current diagnosis of cardiac dysrhythmias or heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, unstable angina requiring medication.
5. Invasive cardiovascular procedure, such as coronary artery bypass graft surgery (CABG), or angioplasty/percutaneous coronary intervention (PCI) within 6 months of screening.
6. History of recurrent severe hypoglycemia (more than 1 event ≤ 6 month)
7. Subjects with clinically active malignancy
8. History of renal disease or abnormal kidney function tests at Screening (glomerular filtration rate [GFR] < 60 mL/min/1.73m2 as estimated using the MDRD equation).
9. History or active hepatic disease or clinically significant abnormal hepatic function tests at Screening suggestive of hepatic impairment (e.g., ALT and/or AST >2 x ULN, GGT >2 x ULN, total bilirubin > 1 x ULN).
10. Subjects with a history or presence of any psychiatric disorder that, in the opinion of the Principal Investigator, might confound the results of the trial or pose additional risk in administering the investigational product to the subject.
11. Personal or family history of hypercoagulability or thromboembolic disease, including deep vein thrombosis and/or pulmonary embolism (PE)
12. History of surgical treatment for obesity (bariatric surgery, gastric banding, etc.) or any other gastrointestinal surgery (including appendectomy, cholecystectomy), any malabsorption disorder, severe gastroparesis, any GI procedure for weight loss (including LAP-BAND®), as well as clinically significant gastrointestinal disorders (e.g. peptic ulcers, severe GERD) at Screening.
13. History of any major surgery within 3 months prior to screening.
14. Any nerve stimulation study or implanted stimulator, including previously or currently implanted vagus nerve stimulator, previously or currently implanted spinal cord stimulator, other implanted electronic medical device, such as implanted pacemaker or cardioverter/ defibrillator (AICD) or history of seizures.
15. Participation in an investigational study within 30 days prior to dosing or 5 half-lives within the last dose of the investigational product given during the investigational study, whichever is longer.
16. Current use of any drugs (other than current treatment for diabetes mellitus) that are known to interfere with glucose or insulin metabolism as stated below in table prohibited medication.
17. Thyroid hormone use is not allowed unless medication is given on a stable dose for at least 3 months prior to screening.
18. Subject is unable to tolerate adhesive tape or has any unresolved adverse skin reaction in the area of the glucose sensor placement.
19. Implanted pacemaker or cardioverter/defibrillator (AICD).
20. History of any active infection, incl. COVID19 (as ruled out by negative PCR test), except mild viral disease, such as common cold, within 30 days prior to screening.
21. Known history or positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2).
22. History of any recent traumatic injury, including intracerebral hemorrhage and visceral injury.
23. Donation or loss of > 500 mL of blood or blood product within 2 months prior to screening.
24. Mental incapacity, unwillingness or language barriers precluding adequate understanding and to follow verbal commands during the ultrasound session or cooperation.
25. An abdominal ultrasound scan or exam within 1 month prior to screening and/or any pre-planned ultrasound examinations during the study, or the need to participate in any unplanned outside ultrasound procedures during study.
26. Use of the agents listed in Prohibited Medications Table below (prescription or nonprescription) is prohibited until completion of all study activities.
27. Identification of risk of hypoglycemia or severely uncontrolled diabetes in screening visit metabolic assessments (CGM, OGTT, and fasting blood draws)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Hepatic Adverse Events - Elevation of liver transaminases AST / ALT. | 2 weeks
  Number of study participants who develop an elevation of liver transaminases compared to baseline parameters, including AST and ALT.
  Grade 1 delta ALT and / or AST <3 x ULN; Grade 2 delta ALT and / or AST >3 - 5 x ULN; Grade 3 delta ALT and / or AST >5 - 20 x ULN; Grade 4 delta ALT and / or AST >20 x ULN.

SECONDARY OUTCOMES:
Number of Metabolism and nutrition disorders - Hypoglycemia | 2 weeks
  Number of study participants who develop Hypoglycemia (- A disorder characterized by laboratory test results that indicate a low concentration of glucose in the blood) after undergoing the study procedure.
  Grade 1 <LLN - 55 mg/dL; <LLN - 3.0 mmol/L Grade 2 <55 - 40 mg/dL; <3.0 - 2.2 mmol/L Grade 3 <40 - 30 mg/dL; <2.2 - 1.7 mmol/L Grade 4 <30 mg/dL; <1.7 mmol/L; Grade 5 life-threatening consequences; seizures Death

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No